CLINICAL TRIAL: NCT06910501
Title: Comparative Effectiveness of Various Educational Approaches on Oral Hygiene in Pediatric Populations
Brief Title: Comparative Effectiveness of Various Educational Approaches on Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilsah Cogulu, Prof.Dr.-Head of Pediatric Dentistry Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ege U. Ethical Com. 21-3.1T/49
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Dental Plaque
MeSH Terms: conditions — Dental Caries; Dental Plaque

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial designed to compare the effectiveness of traditional educational methods and a mobile application (Brush DJ) in promoting oral hygiene habits among healthy children aged 5-12 years.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and the dental professional delivering the interventions were not blinded. However, the examiner (outcomes assessor) conducting clinical assessments was blinded to the intervention groups to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized oral hygiene instruction using a toothbrush and model (Experimental): Traditional Method: Individualized oral hygiene instruction using a toothbrush and model (n=50).
  Interventions: Other: Traditional oral hygiene instruction
- Education through a slide-based PowerPoint presentation (Experimental): Digital Slide-Based Education: Education through a slide-based PowerPoint presentation (n=50).
  Interventions: Other: Digital slide-based education
- Use of the Brush DJ mobile application (Experimental): Mobile Application - Brush DJ: Use of the Brush DJ mobile application, which includes gamified elements such as music, timers, and oral hygiene tips to encourage brushing (n=50).
  Interventions: Other: Brush DJ mobile appliaction

INTERVENTIONS:
Other: Traditional oral hygiene instruction — Individualized demonstration of proper toothbrushing techniques using a toothbrush and a dental model. Conducted by a trained dental professional.
  Arms: Individualized oral hygiene instruction using a toothbrush and model
Other: Digital slide-based education — Educational session using a PowerPoint presentation on a tablet or projector. The session includes visual aids to explain proper brushing techniques, the importance of oral hygiene, and the effects of poor dental care.
  Arms: Education through a slide-based PowerPoint presentation
Other: Brush DJ mobile appliaction — Children use the Brush DJ app, which includes gamified elements such as music, timers, and oral hygiene tips to encourage proper brushing habits. The app provides reminders and engaging content to maintain motivation.
  Arms: Use of the Brush DJ mobile application

SUMMARY:
Background: Dental caries constitutes a major global public health challenge, posing substantial burdens on both oral health outcomes and healthcare systems worldwide, with far-reaching implications for prevention, treatment, and economic resources. Regular tooth brushing is recognized as the most effective preventive measure against dental caries. However, motivating children to adopt and maintain proper oral hygiene behaviors remains a significant challenge. This study aims to evaluate and compare the effectiveness of traditional education methods and a mobile application in promoting oral hygiene habits among children.

Methods: The study included 150 children who attended routine dental examinations. Parents completed a baseline questionnaire to assess their child's oral hygiene habits. Baseline clinical measurements were recorded, including dental caries indices (dft/DMFT, dfs/DMFS), dental plaque, and gingival index scores. Participants were randomly allocated into three groups: Group-1: received individualized oral hygiene instruction using a model and toothbrush; Group-2: received slide-based oral hygiene education; and Group-3: utilized the Brush DJ mobile application. After three months, follow-up assessments were conducted, including a repeated parental questionnaire, clinical evaluations, and a parental satisfaction survey. Statistical analyses were performed using SPSS 25.0 with chi-square, Kruskal-Wallis, and Fisher's Exact tests.

Study Design: This prospective, randomized controlled study compared the effectiveness of traditional educational methods and a mobile application (Brush DJ) in promoting oral hygiene habits among 150 healthy children aged 5-12 years. Ethical approval was obtained from the institutional ethics committee (approval no.: 21-3.1T/49, date: March 18, 2021). Written informed consent was obtained from the parents of all participating children.

Study Population: Participants were recruited from routine dental examinations at Ege University Faculty of Dentistry, Department of Pediatric Dentistry. The sample size was determined through power analysis to ensure statistical significance. Inclusion criteria were children without systemic diseases, no ongoing orthodontic treatment, and willingness to participate. Children with special healthcare needs or those unwilling to participate were excluded.

Baseline Assessments: At baseline, parents completed a structured questionnaire on their child's oral hygiene habits, including frequency and duration of tooth brushing, parental supervision, and fluoride toothpaste use. Clinical oral examinations were conducted under standardized conditions.

The following indices were recorded:

Dental caries indices: dft/DMFT and dfs/DMFS.

Plaque Index (PI): To assess dental plaque presence.

Gingival Index (GI): To evaluate gingival inflammation.

Participants were randomly assigned to one of three groups using block randomization (block size: six):

Group 1: Individualized oral hygiene instruction using a toothbrush and model (n=50).

Group 2: Slide-based education via PowerPoint on a tablet or projector (n=50).

Group 3: Use of the Brush DJ mobile application, incorporating gamification elements such as music, timers, and oral hygiene tips (n=50).

Each intervention was delivered individually to children and their parents by a trained dental professional.

Follow-Up Assessments: After three months, participants attended a recall visit, during which parents completed a follow-up questionnaire. Clinical examinations were repeated to reassess dft/DMFT, dfs/DMFS, plaque index, and gingival index scores.

Parental Satisfaction Survey: Parents evaluated the educational interventions based on ease of use, engagement, and effectiveness in motivating their child. A four-question Likert-scale (1-5 points) parental satisfaction survey was administered.

Statistical Analysis: Data were analyzed using SPSS 25.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics were presented as means ± standard deviations for continuous variables and as frequencies/percentages for categorical variables. The chi-square test, Kruskal-Wallis test, and Fisher's Exact test were used to assess differences between groups. A p-value of <0.05 was considered statistically significant.

DETAILED DESCRIPTION:
Detailed Description:

Study Design This prospective, randomized controlled study was conducted to compare the effectiveness of traditional educational methods and a mobile application (Brush DJ) in promoting oral hygiene habits among 150 (75 girls, 75 boys) healthy children aged 5-12 years. Ethical approval was obtained from the institutional ethics committee prior to the commencement of the study (approval no.: 21-3.1T/49, date: March 18, 2021). Written informed consent was obtained from the parents of all participating children.

Study Population A total of 150 healthy children aged 5-12 years were recruited from those attending routine dental examinations at Ege University Faculty of Dentistry Department of Pediatric Dentistry. The sample size of 150 participants was determined based on a power analysis to ensure adequate statistical power for detecting significant differences between the educational interventions, considering an expected effect size. Inclusion criteria included children with no systemic diseases, no ongoing orthodontic treatment, and patients and their parents willing to participate in the study. Children with special healthcare needs and who did not accept to participate in the study were excluded.

Baseline Assessments At baseline, parents completed an eleven-question structured questionnaire designed to assess their child's oral hygiene habits, including the frequency and duration of tooth brushing, supervision by parents, and use of fluoride toothpaste. Clinical oral examinations were conducted by a single calibrated examiner under standardized conditions.

The following indices were recorded by a calibrated examiner:

Dental caries indices: Decayed, filled, missing teeth (dft/DMFT) and decayed, filled, missing surfaces (dfs/DMFS).

Plaque Index (PI): To assess the presence of dental plaque. Gingival Index (GI): To evaluate gingival inflammation. Participants were randomly assigned to one of the three intervention groups using a computer-generated block randomization method with a fixed block size of six to ensure balanced group allocation throughout the study.

Group 1: Individualized oral hygiene instruction using a toothbrush and model (n=50).

Group 2: Education through a slide-based PowerPoint presentation, delivered on a tablet or projector (n=50).

Group 3: Use of the Brush DJ mobile application, which incorporates gamified elements such as music, timers, and oral hygiene tips to encourage brushing (n=50).

Each intervention was delivered individually to children and their parents by a trained dental professional.

Follow-Up Assessments After three months, participants returned for a recall visit. Parents completed a follow-up questionnaire assessing changes in their child's oral hygiene behaviors. Clinical examinations were repeated to reassess the dental caries indices (dft/DMFT, dfs/DMFS), plaque index, and gingival index.

Parental Satisfaction Survey At the recall visit, parents were asked to complete a satisfaction survey to evaluate their perceptions of the educational interventions, including ease of use, engagement, and effectiveness in motivating their child. The Parental Satisfaction Survey consisting of four questions, scored out of 5 (1-5 points, from "strongly disagree" to "strongly agree") according to Likert scaling was performed on the parents.

Statistical Analysis All data were analyzed using SPSS software version 25.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics were presented as means ± standard deviations for continuous variables and as frequencies and percentages for categorical variables. The chi-square test, Kruskal-Wallis test, and Fisher's Exact test were used to assess differences between groups. A p-value of <0.05 was considered statistically significant." modify this paragraph according to this review: Please remove all information pertaining to the results and conclusions of the study from the record. After the Protocol Section of a record has been registered, results information can be entered in the Results Section of the record by clicking on "Enter Results" on the Record Summary page. Information on how to enter results is provided on the Results Data Entry page (found in the Help menu on the PRS Home page). Please note that any relevant results-related citations can be added to the References module of the record's Protocol Section.

ELIGIBILITY:
Inclusion Criteria:

No systemic diseases No ongoing orthodontic treatment Patients and their parents willing to participate in the study.

Exclusion Criteria:

Children with special healthcare needs Children who did not accept to participate in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Dental plaque index | 3 months
  After three months, participants returned for a recall visit. Clinical examinations were repeated to reassess the plaque index.
  Plaque index 0: No plaque is in the area adjacent to the gingiva.
  Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
  Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
  Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.

SECONDARY OUTCOMES:
Gingival index | 3 months
  After three months, participants returned for a recall visit. Clinical examinations were repeated to reassess the gingival index. Gingival index 0: Healthy gums.
  Gingival index 1: Mild discolouration and oedematous gingiva. No bleeding on probing.
  Gingival index 2: Red, oedematous and shiny gingiva. There is bleeding on probing.
  Gingival index 3: Red, oedematous and ulcerated gingiva. There is spontaneous bleeding.

OTHER OUTCOMES:
Oral hygiene motivation | 3 months
  After three months, participants returned for a recall visit. Parents completed a follow-up questionnaire assessing changes in their child's oral hygiene behaviors.After three months, participants returned for a recall visit. Parents completed a follow-up questionnaire assessing changes in their child's oral hygiene behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) Sharing Statement: De-identified individual participant data (IPD) collected during the study, including questionnaire responses, clinical indices (dft/DMFT, dfs/DMFS, Plaque Index, Gingival Index), and follow-up assessments, will be shared with other researchers upon request.
  Data Availability: The IPD will be made available after publication of the study results, for up to five years.
  Access Criteria: Researchers must submit a formal request outlining the purpose of the data use, and approval will be subject to ethical considerations and institutional guidelines.
  Data Sharing Mechanism: Data will be shared through a secure institutional repository or via direct communication with the principal investigator.
  Restrictions: Personally identifiable information will not be shared, and data use must comply with ethical and legal regulations governing research data privacy.
Supporting Information: Study Protocol
Time Frame: 20 March 2025-